CLINICAL TRIAL: NCT06179901
Title: The Effect of Early MSAT Treatment on Sciatica Caused by Traffic Accidents : A Pragmatic Randomized Controlled Pilot Clinical Trial
Brief Title: The Effect of Early MSAT Treatment on Sciatica Caused by Traffic Accidents.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2023-07
Record Dates: First submitted 2023-11-12; First posted 2023-12-22 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Sciatica; Radiating Pain; Paresthesia; Dysesthesia
Keywords: MSAT; Sciatica; Radiating pain; Paresthesia; Dysesthesia; Acupuncture
MeSH Terms: conditions — Sciatica; Pain; Paresthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrative Korean Medicine Treatment group(IKMT group) (Active Comparator)
  Interventions: Procedure: Integrative Korean Medicine Treatment
- MSAT group (Experimental)
  Interventions: Procedure: Integrative Korean Medicine Treatment; Procedure: lower limb motion style acupuncture treatment

INTERVENTIONS:
Procedure: Integrative Korean Medicine Treatment — acupuncture treatment, chuna, pharmacoacupuncture, Korean herbal medicine, cupping, moxibustion.
Procedure: lower limb motion style acupuncture treatment — Motion Style Acupuncture Treatment(MSAT) is a therapeutic technique using acupuncture needle created in Jaseng Hospital. This treatment involves patients with musculoskeletal pain to move the part of their body actively during acupuncture treatment under physicians' observation.
  Arms: MSAT group

SUMMARY:
The investigators would like to conduct a pilot study prior to a practical randomized control study on the effectiveness of initial MSAT treatment on inpatients complaining of radiating pain and abnormal sensation in the lower extremities caused by traffic accidents.

DETAILED DESCRIPTION:
The stimulation of the nerve roots due to physicochemical causes can lead to symptoms along the distribution area of those nerves, such as radiating pain, numbness, a sensation of heat, dullness in sensation, muscle weakness, and more. While radiating pain and abnormal sensations typically arise from lumbar disc herniation, they can also result from peripheral nerve entrapment, like in radiculopathy. Traditional Korean medicine treatments for radiating pain involve acupuncture, pharmacoacupuncture, moxibustion, cupping and Chuna therapy.

Motion Style Acupuncture Treatment (MSAT) combines traditional acupuncture with neurophysiological theories, focusing on administering acupuncture at the affected area and subsequently involving active or passive movements. Studies have shown the efficacy of MSAT in treating various acute and chronic neuromuscular disorders like low back pain, brachial plexus injury, and temporomandibular joint disorders. Although there have been reports of the effectiveness of pelvic MSAT treatment in patients complaining of lumbar and radiating pain due to lumbar disc herniation, research on the initial effects of MSAT treatment specifically targeting traffic accident victims is still lacking. MSAT has been developed as an emergency acupuncture method that enhances blood circulation by adding movement to traditional acupuncture, offering quick pain relief and restoring range of motion.

Given the significant impact of a traffic accident, positive effects could be anticipated in alleviating radiating pain and restoring reduced range of motion through MSAT, especially when these symptoms arise following such a traumatic event.

ELIGIBILITY:
Inclusion Criteria:

1. a person who has no problem in language communication
2. men and women between the ages of 19 and 69
3. a patient hospitalized for treatment in a car accident
4. A person who complains of radiating pain or abnormal sensation in the lower extremities within three days after a traffic accident
5. A person with a lower extremity radiating pain or abnormal sensation of NRS (Numeric Rating Scale) 5 or higher
6. A person who voluntarily agrees to participate in clinical trials and signs a consent form

Exclusion Criteria:

1. Patient diagnosed with certain serious diseases that may cause radiation pain: malignant tumors, spinal fractures, spinal infections, inflammatory spondylitis, etc
2. Patient with progressive neurological deficits or severe neurological symptoms such as Mami syndrome
3. Patient who has undergone surgery, procedures, or is scheduled to undergo surgery on the lumbar spine or lower extremities within the last 3 weeks
4. Patient with other chronic conditions that may interfere with interpretation of treatment effects or results: cardiovascular disease, kidney disease, active hepatitis, diabetic neuropathy, dementia, severe mental illness, epilepsy, etc
5. Patient who may be inadequate or unsafe with acupuncture treatment: hemorrhagic disease, people on anticoagulant therapy, people with severe cardiovascular disease, pregnancy, and infection Severe diabetic patients, seizure disorders, etc. that are concerned
6. Patient currently taking steroids, immunosuppressants, mental illness medications or other medications that may affect research results
7. Patient Participating in clinical trials other than observational studies without therapeutic intervention
8. Patient who has difficulty filling out consent forms to participate in research
9. Patient deemed difficult to conduct this clinical study when judged by the research director

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-10-06 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale of sciatica(NRS of sciatica) | visit 1 (Admission 1 day), visit 2 (Hospital day 2), visit 3(Hospital day 3), visit 4 (Hospital day 4), visit 5 (Hospital day 5), visit 6 (Discharge 1 day), visit 7 (13 day after admission)
  The degree of radiation pain or abnormal sensation in the patient is evaluated through a numerical pain scale. The numerical pain scale is an index expressed by objectifying the degree of subjective pain into numbers for patients over 12 years of age who can communicate and understand the concept of numbers. The patient's pain level is quantified by zero pain and ten pain that cannot be tolerated as death, and is mild (1-4 points), moderate (5-6 points), and severe (7-10 points).

SECONDARY OUTCOMES:
NRS of Lower back pain(NRS of LBP) | visit 1 (Admission 1 day), visit 2 (Hospital day 2), visit 3(Hospital day 3), visit 4 (Hospital day 4), visit 5 (Hospital day 5), visit 6 (Discharge 1 day), visit 7 (13 day after admission)
  In addition to radiation pain and abnormal sensation, the degree of additional low back pain is evaluated together on a numerical pain scale. Write the degree of pain of the patient by stating that the state without pain at all is 0, and the pain that cannot be tolerated as if dying is 10.
Oswestry disability index(ODI) | visit 1 (Admission 1 day), visit 2 (Hospital day 2), visit 3(Hospital day 3), visit 4 (Hospital day 4), visit 5 (Hospital day 5), visit 6 (Discharge 1 day), visit 7 (13 day after admission)
  It is a questionnaire that measures the discomfort patients feel in their daily lives due to back pain, radiating pain in the lower extremities, and abnormal sensations. It is a functional evaluation tool that measures the availability of 10 daily activity.
European Quality of Life-5 Dimensions(EQ-5D) | visit 1 (Admission 1 day), visit 2 (Hospital day 2), visit 3(Hospital day 3), visit 4 (Hospital day 4), visit 5 (Hospital day 5), visit 6 (Discharge 1 day), visit 7 (13 day after admission)
  EQ-5D is one of the most widely used tools in the health care sector to measure health-related quality of life (HRQOL). It is a questionnaire that evaluates the current HRQOL by dividing it into five categories: mobility (M), self-care (SC), user activity (UA), pain/disability (PD), and anxiety/depression (AD). Each item is evaluated in Phase 1 (no problem at all), Phase 2 (slight problem), Phase 3 (moderate problem), Phase 4 (severe problem), and Phase 5 (severe problem).
  The EQ-5D Index is an index that calculates health status as a quantitative single value by assigning quality weights to each of the five items of EQ-5D. In this study, quality weights for Koreans at the Korea Centers for Disease Control and Prevention are used and calculated as in the formula below.
  EQ-5D Index
  = = 1 - (0.05 + 0.096 × M2 + 0.418 × M3 + 0.046 × SC2 + 0.136 × SC3 + 0.051 × UA2 + 0.208 × UA3 + 0.037 × PD2 + 0.151 × PD3 + 0.043 × AD2 + 0.158 × AD3 + 0.050 × N3)
Patient Global Impression of Change(PGIC) | visit 1 (Admission 1 day), visit 2 (Hospital day 2), visit 3(Hospital day 3), visit 4 (Hospital day 4), visit 5 (Hospital day 5), visit 6 (Discharge 1 day), visit 7 (13 day after admission)
  PGIC is an index that subjectively evaluates the degree of improvement after treatment by patients. The subjective criteria for improvement and deterioration are ambiguous, so it is usually used as a tool to evaluate treatment satisfaction. The criteria can be checked by analyzing changes in pain and dysfunction indicators for patients who are satisfied with treatment.
Straight Leg Raise Test(SLRT) | visit 1 (Admission 1 day), visit 2 (Hospital day 2), visit 3(Hospital day 3), visit 4 (Hospital day 4), visit 5 (Hospital day 5), visit 6 (Discharge 1 day), visit 7 (13 day after admission)
  It is a physical test performed on patients complaining of urticaria and radial pain and is performed in an supine position. The examiner holds the patient's heel with one hand, holds the patient's knee with the other hand, and raises his leg to bend the hip joint while fixing it so that the patient's knee does not bend. Check the angle at which the patient feels uncomfortable with back pain or radiating pain.
  If the knee muscle is a problem when the lower extremity is upright, it is simply related to the back of the thigh, and if the lower extremity radiating pain appears along with nerve driving, it is considered positive. If there is a space-occupying disease such as intervertebral disc hernia, it may indicate back pain or radial pain on the affected side during the tendon examination. Since it is a method of reproducing the patient's pain, the tendon leg is performed first and then the affected leg is examined.
Lumbar Range of motion(Lumbar ROM) | visit 1 (Admission 1 day), visit 2 (Hospital day 2), visit 3(Hospital day 3), visit 4 (Hospital day 4), visit 5 (Hospital day 5), visit 6 (Discharge 1 day), visit 7 (13 day after admission)
  Measure the active range of lumbar flexion, extension, lateral flexion, and rotation. Evaluate whether there is a limitation in the range of motion due to the patient's back pain and radiating pain.
Adverse event(AE) | visit 1 (Admission 1 day), visit 2 (Hospital day 2), visit 3(Hospital day 3), visit 4 (Hospital day 4), visit 5 (Hospital day 5), visit 6 (Discharge 1 day), visit 7 (13 day after admission)
  It refers to undesirable and unintended objective symptoms, subjective symptoms, or diseases that appear after the procedure during the clinical trial process. It is not necessary to have a causal relationship with the procedure. During the study period, it is collected through patient symptom reports and researcher observations, and the causal relationship between the types of adverse reactions and treatment interventions is written on the EMR. Follow-up observation is conducted when an adverse reaction occurs, and if a serious level of adverse reaction is found, report it quickly.
Severity of L-spine HIVD(Herniated intervertebral disc) or lumbar stenosis on MRI | through study completion, an average of 1 month
  Data is collected retrospectively through EMR records for research patients who took L-SPINE MRI. The degree of escape and stenosis of the intervertebral disc on MRI is divided into mild, subtle, moderate, and severe. The stage of intervertebral disc escape is divided into bulding, protusion, extrusion, and sequencing, and the direction of escape is classified into central, subarticular, formal, lateral, and interior. Stenosis will be classified as central, lateral repair, and formal. L-spine MRI is evaluated through retrospective chart review during the study period regardless of the patient's admission and discharge.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, PhD, Study Chair — Bucheon Jaseng Hospital of Korean Medicine
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No